CLINICAL TRIAL: NCT04851847
Title: A Clinical Trial to Evaluate the Safety and Effectiveness of Resorbable Collagen Membrane - MatrixflexTM for the Treatment of Periodontal Intrabony Defects
Brief Title: A Clinical Trial to Evaluate the Safety and Effectiveness of Resorbable Collagen Membrane - MatrixflexTM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Collagen Matrix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D20190472-P
Record Dates: First submitted 2021-04-14; First posted 2021-04-21 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Periodontal Diseases; Intrabony Defects; Guided Tissue Regeneration
Keywords: resorbable collagen membrane
MeSH Terms: conditions — Periodontal Diseases | interventions — Guided Tissue Regeneration

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- MatrixflexTM resorbable collagen membrane (Experimental): Experimental arm using the Matrixflex Resorbable Collagen Membrane for treatment of periodontal intrabony defects
  Interventions: Device: Guided Tissue Regeneration (GTR)
- control group membrane (Active Comparator): Control arm using the Comparator Xenograft Resorbable Collagen Membrane or treatment of periodontal intrabony defects
  Interventions: Device: Guided Tissue Regeneration (GTR)

INTERVENTIONS:
Device: Guided Tissue Regeneration (GTR) — Use of resorbable collagen membrane to treat periodontal intrabony defects.

SUMMARY:
This is a randomized, single blind, parallel-arm, multi-center, non-inferior clinical trial. 174 patients are recruited in total, and they are treated by Guided Tissue Regeneration (GTR). The patients are split in to two groups evenly: 87 in the experimental group and 87 in the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 65 years, male or female;
2. patients were clinically diagnosed with chronic periodontitis according to the international classification of periodontal disease in 1999;
3. Only solitary lesion site requires surgical treatment and must meet the following criteria:

   1. The baseline PD≥7 mm ;
   2. After debridement during operation, the defect of the vertical bone at the adjacent surface ≥4mm, and at least one alveolar buccal wall can be detected;
   3. The wideness of the keratinized gingiva≥2 mm;
   4. Based on the X-Ray image, the dental crowns at the bottom of the bone socket should be at least 3mm;

Exclusion Criteria:

1. The test tooth has open surgical debridement history within the most recent one years;
2. Known allergy to collagen of animal origin;
3. Clinical or radiographic signs of untreated acute infection at the surgical site, apical pathology, root fracture, severe root irregularities, cemental pearls, cemento-enamel projections not easily removed by odontoplasty, untreated carious lesions at the cemento-enamel junction (CEJ) or on the root surface, subgingival restorations and/or restorations with open margins at or below the CEJ;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-07-20 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
The change of CAL at 12 weeks after surgery | 12 weeks
  Assessment of clinical attachment level
The change of CAL at 24 weeks after surgery | 24 weeks
  Assessment of clinical attachment level
The change of PD at 12 weeks after surgery | 12 weeks
  Assessment of Probing Depth
The change of PD at 24 weeks after surgery | 24 weeks
  Assessment of Probing Depth

SECONDARY OUTCOMES:
The ratio between Baseline and gingival recession (GR) at 12 weeks after surgery. | 12 weeks
  Effect on Gingival recession
The ratio between Baseline and gingival recession (GR) at 24 weeks after surgery. | 24 weeks
  Effect on Gingival recession

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Y, Yan F, Chen L, Zhao L, Liu M, Ge S, Chen CY, Kim DM, Shu R. Crosslinked Versus Non-Crosslinked Resorbable Collagen Membranes for Periodontal Regeneration: A Multicenter, Randomized, Double-Blind, Non-Inferiority Clinical Trial. J Periodontal Res. 2025 Jan 12. doi: 10.1111/jre.13382. Online ahead of print. PMID 39799466